CLINICAL TRIAL: NCT02272985
Title: A [15O]H2O PET-CT Pilot Study Comparing Cerebral Blood Flow Before, During and After Hemodialysis
Brief Title: Cerebral Blood Flow During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Principal Investigator, dr. C.F.M. Franssen, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABR 48969
Record Dates: First submitted 2014-10-13; First posted 2014-10-23 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Haemodialysis-induced Symptom
Keywords: cerebral blood flow; hemodialysis
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBF change during hemodialysis (Other): [15O]H2O PET-CT scan and NIRS (Invos)
  Interventions: Other: [15O]H2O PET-CT scan; Other: NIRS (Invos)

INTERVENTIONS:
Other: [15O]H2O PET-CT scan — All participants will undergo 3 [15O]H2O PET-CT scans during the hemodialysis study session
Other: NIRS (Invos) — All participants will undergo near infrared spectroscopy (NIRS) during the hemodialysis study session.

SUMMARY:
The purpose of this study is to evaluate the effect of the hemodialysis procedure on cerebral blood flow (CBF) in elderly maintenance hemodialysis (HD) patients. The investigators hypothesize that HD induced blood pressure changes are associated with a fall in global and/or regional CBF during HD. Second, the investigators hypothesize that near infrared spectroscopy (NIRS) will correlate with CBF measured by[15O]H2O PET.

DETAILED DESCRIPTION:
The investigators aim to include 14 participants. Each participant will undergo a single HD study session in the PET center of the UMCG. During this study session, each participant will undergo three gated [15O]H2O PET-CT scans before, during (after 20 minutes) and at the end of the HD session. NIRS will be used to measure cerebral tissue regional oxygen saturation (rSO2) during the HD study session. INVOS (In Vivo Optical Spectroscopy), a monitoring device, will be used to measure rSO2, with sensors placed bilaterally on the patient forehead. Participants will further undergo a MRI scan of the brain, bilateral carotid artery duplex echosonography, cognitive testing, blood pressure and heart rate measurements during the HD study session, and laboratory measurements during the HD study session.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥ 65 years, HD patients who have been treated with maintenance HD, of which at least 6 patients for a longer period of time (>1 year).
* Patients must have an arteriovenous fistula without recirculation
* The hemoglobin value must be in the target range (6.2 - 8mmol/l) since at least 1 month

Exclusion Criteria:

* The absence of informed consent
* Diagnosis of dementia, hydrocephalus, history of raised intracranial pressure, significant (>70%) carotid artery stenosis, end-stage liver disease.
* Actively treated cancer
* Actual hospital admission at timing of HD study session
* MRI incompatible implants in the body or any other contraindication for MRI
* Claustrophobia
* The refusal to be informed of significant carotid artery stenosis or structural brain abnormalities that could be detected during the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casper FM Franssen, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- CBF Change: Hemodialysis patients that underwent 3 PET-scans during a hemodialysis study-session.
Period: Overall Study
Arm/Group | CBF Change
Started | 15
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — hip fracture | 1
Not completed — kidney transplantation | 1

BASELINE CHARACTERISTICS:
Groups:
- CBF Change During HD: Arm/Group is not applicable.
Arm/Group | CBF Change During HD
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 15
dialysis vintage [Median (Full Range); unit: months] — Population: Three patients withdrew their consent before the actual start of the study. Therefore, we did not include them in the analyses.
  months
    number analyzed (Participants) | 12
    (all) | 47 [11 to 319]
diabetes [Count of Participants; unit: Participants] — Population: Three patients withdrew their consent before the actual start of the study. Therefore, we did not include them in the analyses.
  Participants
    number analyzed (Participants) | 12
    (all) | 3
hypertension [Count of Participants; unit: Participants] — Population: Three patients withdrew their consent before the actual start of the study. Therefore, we did not include them in the analyses.
  Participants
    number analyzed (Participants) | 12
    (all) | 11
heart failure [Count of Participants; unit: Participants] — Population: Three patients withdrew their consent before the actual start of the study. Therefore, we did not include them in the analyses.
  Participants
    number analyzed (Participants) | 12
    (all) | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in CBF From Baseline (Before Start of the Hemodialysis Study Session), at 20 Minutes, and at the End of the Hemodialysis Study Session, Measured by [15O]H2OPET-CT
Time Frame: at t= -5 minutes, t= 20 minutes, and at t=220 minutes.The change from baseline (-5min) to the end of hemodialysis (220min) is reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/100g/min
Groups:
- Global CBF Change During HD: All patients (n=12)
Arm/Group | Global CBF Change During HD
Number analyzed (Participants) | 12
mL/100g/min | -4.1 [-7.3 to -0.9]
Statistical Analysis 1: Comparison: Global CBF Change During HD; Test type: Other; p = 0.03, Mixed Models Analysis — the p value was calculated

2. Secondary Outcome: Change in rSO2 From Baseline (Before Start of the Hemodialysis Study Session), at 20 Minutes, and at the End of the Hemodialysis Study Session, Measured by NIRS
Description: Change in rSO2, between baseline (-5 minutes) and the end of the hemodialysis (t=220 minutes) study session.
Time Frame: at t= -5 minutes, t= 20 minutes, and at t=220 minutes.The start of dialysis was considered as t=0. Therefore, baseline is t=-5minutes.
Measure: Mean (95% Confidence Interval); unit: percentage of regional oxygen saturation
Groups:
- rSO2 Change During Hemodialysis: [15O]H2O PET-CT scan and NIRS (Invos)
  [15O]H2O PET-CT scan: All participants will undergo 3 [15O]H2O PET-CT scans during the hemodialysis study session
  NIRS (Invos): All participants will undergo near infrared spectroscopy (NIRS) during the hemodialysis study session.
Arm/Group | rSO2 Change During Hemodialysis
Number analyzed (Participants) | 12
percentage of regional oxygen saturation
  Left rSO2 | -4.2 [-6.6 to -1.8]
  Right rSO2 | -3.1 [-6.4 to 0.3]
Statistical Analysis 1: Comparison: rSO2 Change During Hemodialysis; Left frontal gray matter:; Test type: Other; p = 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: rSO2 Change During Hemodialysis; Right frontal gray matter:; Test type: Other; p = 0.08, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | CBF Change During HD
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBF Change During HD (N=15)
dialysis hypotension (Vascular disorders) | 1 (1) — The patient experienced dialysis hypotension at the end of the hemodialysis session. This patient had a history of dialysis hypotension episodes. He made an uneventful recovery.
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — The patient experienced a hip fracture just after signing informed consent but before the study was started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No